CLINICAL TRIAL: NCT04195451
Title: RE-ENERGIZE FONTAN: A RandomizEd Exercise INtERvention DesiGned to MaximIZE Fitness in Pediatric FONTAN Patients
Brief Title: Re-Energize Fontan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: The Methodist Hospital Research Institute (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Seda Tierney, Associate Professor, Pediatrics, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 46606; R33HL146775 (NIH); 1R61HL146775-01A1 (NIH)
Record Dates: First submitted 2019-12-06; First posted 2019-12-11 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Single-ventricle
Keywords: Fontan palliation
MeSH Terms: conditions — Univentricular Heart

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Live Video-Supervised Exercise Intervention Arm (Experimental): Patients randomized to exercise intervention at baseline will participate in live-video-supervised exercise sessions x3/week for 3 months, and then will follow a maintenance regimen for 6 months. During maintenance, patients will continue live-video-supervised exercise sessions, only x1/week, and will be instructed to exercise on their own x2/week following an individualized prescribed exercise program and use their heart rate monitor as an activity tracker.
  Interventions: Other: Live-Video-Supervised Exercise Intervention
- Live-Video-Supervised Exercise Control Arm (Experimental): Patients randomized to usual care at baseline will receive usual care for 9 months and will then start the 3-month exercise intervention of live-video-supervised exercise sessions x3/week for 3 months.
  Interventions: Other: Usual Care then Live-Video Supervised Exercise Intervention

INTERVENTIONS:
Other: Live-Video-Supervised Exercise Intervention — The live-video-supervised exercise intervention includes exercise sessions x3/week for 3 months, and then maintenance regimen for 6 months. Maintenance includes live-video-supervised exercise sessions, only x1/week, and self-exercise x2/week following an individualized prescribed exercise program and use their heart rate monitor as an activity tracker.
  Arms: Live Video-Supervised Exercise Intervention Arm
Other: Usual Care then Live-Video Supervised Exercise Intervention — Patients randomized to usual care at baseline will receive usual care for 9 months and will then start the live-video-supervised exercise intervention that includes exercise sessions x3/week for 3 months.
  Arms: Live-Video-Supervised Exercise Control Arm

SUMMARY:
Survival of children with single ventricles ("half a heart") beyond the neonatal period has increased dramatically with the staged Fontan palliation. Yet, long-term morbidity remains high. By the age of 40, 50% of Fontan patients will have died or undergone heart transplantation. With >1,000 Fontan palliations performed in the US annually, there is a burgeoning population of Fontan patients at risk for progressive heart failure and death. Factors that contribute to onset and progression of heart failure in Fontan patients remain incompletely understood. However, it is established that Fontan patients have poor exercise capacity, associated with a greater risk of morbidity and mortality, in addition to decreased muscle mass, abnormal muscle function, and endothelial dysfunction contributing to disease progression. In adult patients with two ventricles and heart failure, reduced exercise capacity, muscle mass, and muscle strength are powerful predictors of poor outcomes, and exercise interventions can not only improve exercise capacity and muscle mass, but also reverse endothelial dysfunction. Limited exercise interventions in children with congenital heart disease have demonstrated that exercise is safe and effective; however, these studies have been conducted in small, heterogeneous groups, and most had few Fontan patients. Furthermore, none of these interventions have studied the impact of exercise on muscle mass or mitochondrial function, or endothelial function. The investigators propose a milestone-driven, randomized controlled trial in pediatric Fontan patients to test the hypothesis that a live-video-supervised exercise (aerobic + resistance) intervention will improve cardiac and physical capacity; muscle mass, strength and function; and endothelial function. The investigators' ultimate goal is the translation of this model to clinical application as an "exercise prescription" to intervene early in pediatric Fontan patients and decrease long-term morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* 8-19 years of age
* Fontan palliation
* Ability to fast overnight
* Cardiac clearance to exercise by primary cardiologist
* Presence of an adult at home during exercise sessions for patients <14 years old
* English-speaking patient.

Exclusion Criteria:

* NYHA Class IV (severe heart failure)
* Acute illness within the past three months
* Active protein losing enteropathy (albumin <2.5 mg/dL)
* Implanted pacemaker
* Cognitive delay deemed severe enough to inhibit the ability to follow the exercise

Ages: 8 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-08-06 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in volume of Oxygen Consumed at Maximal Exertion | Baseline, 3 months, 9 months, 12 months
  In Fontan patients, peak VO2 is a powerful predictor of poor outcomes. The subjects will undergo progressive cardiopulmonary exercise testing with continuous monitoring by 12-lead EKG and gas exchange by measuring breath-to-breath ventilation. Exercise capacity will be measured by a cardiopulmonary exercise test to obtain the peak VO2

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Lucile Packard Children Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gallegos FN, Bernstein D, Punn R, Long J, Stauffer KJ, Thorson K, Chen S, Lui MC, Olson I, Myers J, Palaniappan L, Tierney S. Systolic performance of the single ventricle, exercise capacity, and endothelial function in pediatric Fontan patients. Am Heart J. 2025 Dec;290:58-68. doi: 10.1016/j.ahj.2025.05.015. Epub 2025 May 31. PMID 40456431
- [Derived] Selamet Tierney ES, Palaniappan L, Leonard M, Long J, Myers J, Davila T, Lui MC, Kogan F, Olson I, Punn R, Desai M, Schneider LM, Wang CH, Cooke JP, Bernstein D. Design and rationale of re-energize fontan: Randomized exercise intervention designed to maximize fitness in fontan patients. Am Heart J. 2023 May;259:68-78. doi: 10.1016/j.ahj.2023.02.006. Epub 2023 Feb 14. PMID 36796574